CLINICAL TRIAL: NCT06257199
Title: Real-Time Morphometric Changes of Temperature-Sensitive NiTi Endodontic Instruments in Relation to Intracanal Temperature
Brief Title: Real-time Measurement of Intra-canal Temperature in Vivo
Status: Completed | Type: Observational
Sponsor: King Abdullah University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20230248
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Healthy Patients
Keywords: Irrigation; Intracanal; temperature

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Included patients will be attending the dental clinics for a root canal treatment. After explaining the procedure and obtaining their consent, the intracanal temperature of the treated tooth will be measured after irrigation with normal saline at 2 different temperatures: 22- and 45-degree Celsius. The intraoral temperature will be recorded using a thermocouple probe inserted inside the canal at the mid-root level. Intraoral temperature will be recorded at the same time using another probe attached to the lingual mucosa. A video will be recorded for the temperature changes over 180 seconds duration starting from the time of placing the irrigation solution into the canal.

DETAILED DESCRIPTION:
- Measurement of intracanal temperature in vivo Healthy patients attending the dental clinics for non-surgical root canal treatment of permanent mandibular first molars will be included in the study after obtaining ethical approval (IRB ethical approval ref. 10/158/2023). Their body temperature will be measured using a non-contact thermometer pointed at the forehead. Any patient with a body temperature higher than 37°C will not be included. The participants will sign a consent form after the procedure is fully explained. Upon rubber dam isolation, access cavity preparation will be performed, and canals will be chemo-mechanically prepared using a ProTaper Gold NiTi rotary system (Dentsply Sirona, Switzerland). Distal canals will be prepared up to the F3.

A four-channel portable thermometer will be used with two K-type thermocouple probes to simultaneously measure both intracanal and intraoral temperatures. The intraoral temperature will be measured by securing the probe in direct contact with the lingual alveolar mucosa under the rubber dam. The intracanal temperature will be measured by another probe inserted inside the distal canal at the mid-root level. The insertion depth will be verified using a preoperative radiograph and a rubber stop. If the probe insertion to that depth is not possible, the tooth will be excluded. Based on a previous study, 20 teeth will be included in the experiment. In each canal, two measurements will be obtained; the first one will be irrigated using a normal saline set at room temperature (RT), and the other measurement will be taken after irrigation using heated temperature (HT) normal saline . The RT irrigation solution will be used while maintaining the ambient temperature of the air-conditioned clinic fixed at 22°C. The HT irrigation solution will be heated using a chairside dental composite heater set at 45°C. The preset temperatures of each irrigation group will be confirmed with 3 repeated measurements.

After securing the thermocouple probe inside the canal, the RT irrigation solution will be applied using a gauge-27 side vented needle. A video camera will be used for recording the change of both intraoral and intracanal temperatures appearing on the digital display of the thermometer for 180 seconds. After 5 min, the canal will be dried, and the HT irrigation solution will be applied repeating the same steps.

The thermocouple probes will be chemically sterilized before each use. From the video recordings, still frames will be extracted at 5-second intervals using the VLC media player plotting the body and intracanal temperature at each time point.

ELIGIBILITY:
Inclusion Criteria:

- Health patients ASA I-II non pregnant women

Exclusion Criteria:

* ASA III and above pregnant women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: health patient attend the Dental teaching center at Jordan university of science and technology were recruited for the current study, patient was aware of the process and signed informed consent in which accept to measure the temperature of the canals, patient was informed with all safty measure.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2024-01-28 (Actual)

PRIMARY OUTCOMES:
Real-time intra canal temperature measurements | 6 months
  assessing the temperature changes inside the root canal system that might influence the rotary files performance

CONTACTS AND LOCATIONS:
Locations (1):
- Dr.Taher Al Omari, Irbid, Jordan